CLINICAL TRIAL: NCT00405158
Title: A RCT in Sweden of Acupuncture and Care Interventions for the Relief of Inflammatory Symptoms of the Breast During Lactation
Brief Title: Study of Acupuncture and Care Interventions for the Treatment of Breast Inflammation During Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karlstad University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 84839
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Mastitis
Keywords: Lactation mastitis; Breast inflammation; Breastfeeding; Care interventions; Acupuncture treatment; Antibiotic therapy
MeSH Terms: conditions — Mastitis; Breast Feeding | interventions — Acupuncture Therapy; Acetaminophen; Cefadroxil; Penicillins; Floxacillin

INTERVENTIONS:
Procedure: Acupuncture treatment
Procedure: Administration of oxytocin nasal spray
Procedure: Improved breast milk removal
Procedure: Warmth applied to breasts
Procedure: Breast massage
Drug: Anti-pyretic medication, paracetamol
Drug: cefadroxil
Drug: penicillin
Drug: flucloxacillin

SUMMARY:
The objective of the study was to test the hypothesis that acupuncture treatment hastens recovery time from inflammatory symptoms of the breast during breastfeeding. 205 mothers with 210 cases of breast inflammation (commonly called "mastitis") during breastfeeding were randomly assigned to one of three treatment groups. There were two groups where acupuncture was used and one without acupuncture. The mothers symptoms were recorded at the onset of health care contact and daily until recovery. All care interventions given, including antibiotic therapy, were monitored. Women who participated were asked to leave a breast milk sample to test for bacterial growth. It was found that acupuncture did not shorten the women's contacts with health care services but did improve their symptoms on contact days 3 and 4. It was seen in this study that only 15 % of women were prescribed antibiotics which was a very low rate of prescription compared to USA, Canada, Australia, Turkey and New Zealand where up to 100% are given antibiotics. Seven women (3.3% of those in the study) developed a breast boil and this is a similar number to a study in Australia where many more were treated by antibiotics. This could mean that many women throughout the world are given antibiotics when in fact they may recover without them. This is an important finding in relation to the fight against antibiotic resistant bacteria.

DETAILED DESCRIPTION:
Objectives: to further compare acupuncture treatment and care interventions for the relief of inflammatory symptoms of the breast during lactation and to investigate the relationship between bacteria in the breast milk and clinical signs and symptoms.

Design: randomised, non-blinded, controlled trial of acupuncture and care interventions.

Setting: a midwife-led breast-feeding clinic in Sweden.

Participants: 205 mothers with 210 cases of inflammatory symptoms of the breast during lactation agreed to participate. The mothers were randomly assigned to one of three treatment groups, two of which included acupuncture amongst the care interventions and one without acupuncture. All groups were given essential care. Protocols, which included scales for erythema, breast tension and pain, were maintained for each day of contact with the breast-feeding clinic. A Severity Index (SI) for each mother and each day was created by adding together the scores on the erythema, breast tension and pain scales. The range of the SI was 0 (least severe) to 19 (most severe).

Findings: There was no significant difference in numbers of mothers in the treatment groups with the lowest possible score for severity of symptoms on contact days 3, 4 or 5. There were no statistically significant differences between the treatment groups for number of contact days needed until the mother felt well enough to discontinue contact with the breast-feeding clinic or for number of mothers prescribed antibiotics. There were significant differences in the mean SI scores on contact days 3 and 4 between the non-acupuncture group and the two acupuncture groups. Mothers with less favourable outcomes (≥ 6 contact days, n = 61) were, at first contact with the midwife more often given advice on correction of the baby's attachment to the breast. An obstetrician was called to examine 20 % of the mothers and antibiotic therapy was prescribed for 15 % of the study population. The presence of Group B streptococci in the breast milk was related to less favourable outcomes.

Key conclusions and implications for practice: If acupuncture treatment is acceptable to the mother, this, together with care interventions such as correction of breast-feeding position and babies' attachment to the breast might be a more expedient and less invasive choice of treatment than the use of oxytocin nasal spray. Midwives, nurses or medical practitioners with specialist competence in breast feeding should be the primary care providers for mothers with inflammatory symptoms of the breast during lactation. The use of antibiotics for inflammatory symptoms of the breast should be closely monitored in order to help the global community reduce resistance development among bacterial pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Lactating mothers with symptoms of breast inflammation
* Any mixture of increased breast tension, fever, breast erythema, lumps in the breast

Exclusion Criteria:

* Non-Swedish speaking
* Psychiatric illness
* Hemorrhagic disease
* Prosthetic heart valves
* Skin infections
* Hepatitis B
* HIV positive.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210
Dates: Start 2002-01; Study Completion 2004-03

PRIMARY OUTCOMES:
Proportion of women with lowest possible scores for symptom severity on days 3,4 and 5 in the three groups
Comparison of the three groups for mean scores for symptom severity on days 3,4 and 5
Comparison of the three treatment groups for number of contact days with health care services until recovery
Proportion of mothers in the three groups with less favourable outcomes (6 or more contact days to recovery)
Comparison of the three groups for proportions of women prescribed antibiotics
Comparison of the three groups for proportions of mothers who developed breast abscess
Proportions of women in the three groups who experienced residual symptoms within 6 weeks which required renewed health care contact
Comparison of the three groups for care interventions used

SECONDARY OUTCOMES:
Amounts of bacteria in the breast milk and correlated to erythema, increased breast tension and pain at first contact
Type of bacteria in breast milk related to favourable outcomes (5 or less contact days) and less favorable outcomes (6 or more contact days)
Differences in care interventions used in relation to favourable/less favourable outcomes
Relationship between the occurrence of residual symptoms and the use of antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Kvist, PhD, Principal Investigator — Karlstads University; Bodil Wilde Larsson, PhD, Study Director — Karlstad University
Locations (1):
- Dept Obstetrics & Gynecology, Helsingborg Hospital, Helsingborg, Skåne County, Sweden

REFERENCES:
- [Background] Kvist LJ, Hall-Lord ML, Rydhstroem H, Larsson BW. A randomised-controlled trial in Sweden of acupuncture and care interventions for the relief of inflammatory symptoms of the breast during lactation. Midwifery. 2007 Jun;23(2):184-95. doi: 10.1016/j.midw.2006.02.003. Epub 2006 Oct 18. PMID 17052823
- See also: Karlstad University Webb page — http://www.kau.se